CLINICAL TRIAL: NCT03158376
Title: Perioperative Gabapentin for Chronic Post-thoracotomy Pain: a Randomized, Double Blind, Placebo-controlled Study.
Brief Title: Preoperative Gabapentin for Chronic Pain After Thoracotomy (GABATHOMIE).
Acronym: GABATHOMIE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: University of Lille Nord de France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014_12; 2014-005226-35 (EudraCT Number)
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Postoperative Pain; Chronic Pain
Keywords: gabapentin; thoracotomy; chronic post-thoracotomy pain; acute post-thoracotomy pain; quality of life; neuropathic pain
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain; Neuralgia | interventions — Gabapentin; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- gabapentin group (Experimental): * the day before surgery : gabapentin 400 mg orally
  * preoperatively (2 hours before surgery) : 3 capsules each containing 400 mg gabapentin (total gabapentin dose 1200 mg) and intravenous infusion of 50 ml of normal saline solution
  * postoperative day 1 to 10 : 400 mg x 3 ( gabapentin 1200 mg daily)
  Interventions: Drug: Gabapentin
- placebo group (Placebo Comparator): * The day before surgery: 1 placebo capsule orally
  * preoperatively (2 hours before surgery) : 3 placebo capsules and intravenous infusion of 75 mg hydroxyzine
  * postoperative day 1 to 10: 1 placebo capsule x 3
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin
  Other Names: gabapentin Biogaran 400 mg capsule
  Arms: gabapentin group
Drug: Placebo
  Other Names: placebo oral capsule (lactose)
  Arms: placebo group

SUMMARY:
To assess the effects of prolonged preoperative gabapentin treatment (10 days) on chronic pain after thoracotomy.

DETAILED DESCRIPTION:
Randomized, double blind study enrolling 200 adults undergoing thoracotomy. Patients receive either 75 mg hydroxyzine before surgery and placebo 3 times daily for 10 days or 1200 mg gabapentin before surgery continued for 10 days. All patients receive also a thoracic epidural analgesia.

Assessment of chronic pain at 3 month with an evaluation by a physician (pain intensity, pain quality and analgesia requirement).

Assessment of acute pain in the early postoperative period (pain intensity, pain quality and analgesia requirement).

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* elective lung resection via thoracotomy

Exclusion Criteria:

* extended pleurectomy and chest wall resection
* previous ipsilateral thoracotomy
* previous ipsilateral radiotherapy
* thoracotomy for pyothorax
* chest injury
* palliative surgery
* contraindicated placement of a thoracic epidural catheter
* allergy to medications on protocol
* pre-existing pain syndrome
* current treatment with morphine, gabapentin, pregabalin, anticonvulsivants or tricyclic antidepressants
* a history of past or current drug addiction
* severe hepatic, renal or cardiovascular disorders
* inability to understand the study protocol or to answer the questionnaires on pain and quality of life
* severe psychiatric disorders
* incompetent adults under some form of guardianship
* refusal of the protocol
* persons without social security coverage
* pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2019-05-24 (Actual)

PRIMARY OUTCOMES:
Persistent chronic post-thoracotomy pain | 3 months after surgery
  Pain intensity is measured on a 11-point numeric pain rating scale ; a score >=0 is considered as chronic pain.

SECONDARY OUTCOMES:
Quantitative pain assessment: Acute postoperative pain intensity | Within the first 10 postoperative days
  Measured on a 11-point numeric rating scale
Quantitative pain assessment: Rescue analgesics requirement | Within the first 3 months after surgery
  consumption of additional analgesics (opioids, nefopam or non steroidal anti-inflammatory drug) and time to first request.
Quantitative pain assessment: volume of epidural infusion | Within the 5 postoperative days
  total dose of epidural local anesthetic and epidural morphine
Qualitative pain assessment: incidence of neuropathic pain | postoperative day 2
  Assessed by DN4 (Neuropathic pain 4), NPSI (Neuropathic Pain Symptom Inventory) and QDSA ( Saint Antoine French questionnaire = McGill questionnaire)
Qualitative pain assessment: incidence of neuropathic pain | postoperative day 6
  Assessed by DN4 (Neuropathic pain 4), NPSI (Neuropathic Pain Symptom Inventory) and QDSA ( Saint Antoine French questionnaire = McGill questionnaire)
Qualitative pain assessment: incidence of neuropathic pain | 3 months after surgery
  Assessed by DN4 (Neuropathic pain 4), NPSI (Neuropathic Pain Symptom Inventory) and QDSA ( Saint Antoine French questionnaire = McGill questionnaire)
Qualitative pain assessment: Rescue analgesics requirement for neuropathic pain | within the first 3 months after surgery
  Time to first request and consumption (doses and length of treatment) of gapapentinoids, amitriptyline
Qualitative pain assessment: Objective assessment of hyperalgesia by the Von Frey filaments test | 3 months after surgery
  60 and 300 g Von Frey filaments test on the thoracotomy area
Heath related quality of life | 3 months after surgery
  measured by EQ-5D-5L questionnaire
Assessment of sedation in the operating room | baseline
  measured by MOAA/S scale ( Modified Observer's Assessment of alternes/sedation Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Desbordes, MD, Principal Investigator — Lille University Hospital
Locations (1):
- Department of Thoracic Surgery, Lille University Hospital, Lille, France

IPD SHARING:
Plan to Share IPD: No